CLINICAL TRIAL: NCT02236156
Title: A Phase 3, Double-blind, Multicentre, Randomised, Placebo-controlled Study to Determine the Efficacy and Safety of SPL7013 Gel to Prevent the Recurrence of Bacterial Vaginosis.
Brief Title: Efficacy and Safety Study of SPL7013 Gel to Prevent the Recurrence of Bacterial Vaginosis (BV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPL7013-018
Record Dates: First submitted 2014-09-05; First posted 2014-09-10 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole; astodrimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1% SPL7013 Gel (Experimental): Inserted in to the vagina on alternate days (i.e. every other day) for 16 weeks
  Interventions: Drug: Metronidazole oral tablets 500mg; Drug: 1% SPL7013 Gel
- Placebo Gel (Placebo Comparator): Inserted in to the vagina on alternate days (i.e. every other day) for 16 weeks
  Interventions: Drug: Metronidazole oral tablets 500mg; Drug: Placebo gel

INTERVENTIONS:
Drug: Metronidazole oral tablets 500mg — One tablet taken orally twice daily for seven consecutive days
Drug: 1% SPL7013 Gel — 5g inserted in to the vaginal on alternate days (i.e. every other day) for 16 consecutive weeks.
  Other Names: VivaGel; astodimer sodium
  Arms: 1% SPL7013 Gel
Drug: Placebo gel — 5g inserted in to the vagina on alternate days (i.e. every other day) for 16 consecutive weeks
  Arms: Placebo Gel

SUMMARY:
A double-blind, phase 3 study to determine the efficacy of SPL7013 Gel when administered on alternate days for 16 weeks, compared to placebo gel in preventing the recurrence of BV in women with a history of recurrent BV.

DETAILED DESCRIPTION:
Eligible participants, with both a history of recurrent BV and a current episode of BV, will receive a seven-day course of oral metronidazole. Participants who are successfully treated for their BV, and continue to be eligible, will be randomly assigned to receive either 1% SPL7013 Gel or placebo gel on alternate days at bed-time for 16 consecutive weeks.

The primary endpoint will be determined at the conclusion of this 16 week treatment phase.

Participants who experience a BV recurrence will be considered to have completed the study. Such participants will receive BV treatment in line with local practice and will not attend any further study visits.

Participants who successfully reach Week 16 without a BV recurrence will enter a 12-week follow-up phase to Week 28.

Participants will attend a study visit at 4-weekly intervals throughout the duration of the study to Week 28 (or up to the point of BV recurrence) to assess recurrence of BV and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Current active episode of BV (diagnosis defined as: at least 3 Amsel criteria; Nugent score of at least 4; presence of BV-related symptoms)
* History of recurrent BV (at least 3 episodes in previous year including current episode)
* Using an effective method of contraception

Exclusion Criteria:

* Test positive for a sexually transmitted infection
* Presence of genital Herpes Simplex Virus (HSV) lesions or Human Papilloma Virus (HPV) lesions requiring treatment
* Abnormal pelvic exam, including presence of other vaginal or urinary tract infections
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 637 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Recurrence of BV where a diagnosis of BV is defined as the presence of at least 3 clinical findings | At or by the Week 16 visit
  Number of participants with a recurrence

SECONDARY OUTCOMES:
Time to recurrence of BV according to the primary efficacy endpoint definition | At or by the Week 28 visit
  Time (days)
Presence of patient-reported BV symptoms | At or by the Week 16 visit
  Number of participants with symptoms
Recurrence of individual Amsel criteria | At or by the Week 16 visit
  Individual Amsel criteria are:
  i) Presence of homogenous vaginal discharge characteristic of BV
  ii) Positive whiff test
  iii) Clue cells representing at least 20% of total epithelial cells
  iv) vaginal fluid pH greater than 4.5
Recurrence of BV as determined by presence of a Nugent score of 7-10 | At or by the Week 16 visit
  Number of participants with a recurrence
Recurrence of BV according to the primary efficacy endpoint definition | At or by the Week 20, 24 and 28 visits
  Number of participants with a recurrence
Recurrence of BV according to the composite definition of at least 3 clinical findings and a Nugent score of at least 4 | At or by the Week 16 visit
  Number of participants with a recurrence
Adverse events (AEs) | Study duration
  Number of participants
Responses to Quality of Life (QoL) Questionnaires | Screening to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Paull, PhD., Study Chair — Starpharma Pty Ltd
Locations (30):
- United States (4):
  - Precision Trials, LLC, Phoenix, Arizona
  - Medical Center for Clinical Research, San Diego, California
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
- Bulgaria (4):
  - Sites Various, Pleven
  - Sites Various, Plovidiv
  - Sites Various, Sofia
  - Sites Various, Stara Zagora
- Czechia (6):
  - Sites Various, Brno
  - Sites Various, České Budějovice
  - Sites Various, Olomouc
  - Sites Various, Písek
  - Sites Various, Prague
  - Sites Various, Vsetín
- Hungary (8):
  - Sites Various, Baja
  - Sites Various, Balatonfüred
  - Sites Various, Budapest
  - Sites Various, Debrecen
  - Sites Various, Gyömrő
  - Sites Various, Komárom
  - Sites Various, Létavértes
  - Sites Various, Zalaegerszeg
- Ukraine (3):
  - Sites Various, Ivano-Frankivsk
  - Sites Various, Kyiv
  - Sites Various, Zaporizhzhia
- United Kingdom (5):
  - Sites Various, Birmingham
  - Sites Various, Coventry
  - Sites Various, Leeds
  - Sites Various, London
  - Sites Various, Plymouth